CLINICAL TRIAL: NCT04409704
Title: Repetitive Transcranial Magnetic Stimulation of the Dorsomedial Prefrontal Cortex as a Treatment for Anorexia Nervosa and Bulimia Nervosa: An Open-Label Case Series
Brief Title: Repetitive Transcranial Magnetic Stimulation of the DMPFC for Anorexia and Bulimia: an Open-Label Case Series
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Klarman Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0771
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Bulimia Nervosa; Anorexia Nervosa
Keywords: Eating Disorders; rTMS; Anorexia; Bulimia
MeSH Terms: conditions — Bulimia Nervosa; Anorexia Nervosa; Feeding and Eating Disorders; Anorexia; Bulimia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 10 Hz (Experimental): 10 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, once daily, 5 days per week for 4-6 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — 10 Hz repetitive transcranial magnetic stimulation to dorsomedial prefrontal cortex, once daily, 5 days per week, 20-30 sessions.
  Other Names: High-frequency rTMS; Magventure DB80 Coil

SUMMARY:
This project proposes to perform a pilot study of fMRI targeted Dorsomedial Prefrontal Cortex repetitive transcranial magnetic stimulation (DMPFC-rTMS) on individuals diagnosed with Bulimia Nervosa (BN) and Anorexia Nervosa (AN). The DMFPC is a novel target for rTMS, is heavily implicated in the regulation of mood and affect, and has been suggested to be involved in AN, BN, major depression, OCD, and PTSD. Improved function in this area might lead to reduced AN and BN symptoms, such as bingeing, purging, and over-activity, perhaps by improved regulation of mood and affect. Improvements in important areas of comorbidity might allow for better response to intensive treatment for AN and BN, and reduce relapse rates after such treatment. The DMPFC may be a more appropriate target for compared to the Dorsolateral Prefrontal Cortex (DLPFC), which has typically been the focus of stimulation in the past. Our initial preliminary pilot work has noted unexpected and significant improvements in some core ED symptoms (bingeing and purging) and in important areas of comorbidity (OCD and PTSD), along with expected improvements in mood. These changes have allowed some treatment resistant patients to either complete intensive treatment or be successful in maintaining their progress post intensive treatment. Subjects will receive up to 30 sessions of bilateral DMPFC-rTMS. Response will be evaluated clinically, via psychometric measures, and pre and post fMRI.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

* Are voluntary and competent to consent to treatment.
* Have met DSM-5 diagnostic criteria for Anorexia Nervosa or Bulimia Nervosa, over the last 6 months at minimum

Exclusion Criteria:

Patients will be excluded if they have:

1. Past or current neurological illness
2. Comorbid schizophrenia
3. Current suicidal intent or plan
4. Contraindications to MRI or rTMS (e.g., metallic implants/foreign bodies)
5. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12-11 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination (EDE) | Change from baseline to 1 week post-treatment completion.
  Weekly Binge/Purge Frequency on Eating Disorder Examination (EDE), a semi-structured interview assessing the full range of the specific psychopathology of eating disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Downar, MD, Principal Investigator — University Health Network, Toronto; Blake Woodside, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodside DB, Dunlop K, Sathi C, Lam E, McDonald B, Downar J. A pilot trial of repetitive transcranial magnetic stimulation of the dorsomedial prefrontal cortex in anorexia nervosa: resting fMRI correlates of response. J Eat Disord. 2021 Apr 17;9(1):52. doi: 10.1186/s40337-021-00411-x. PMID 33865456